CLINICAL TRIAL: NCT07120256
Title: Different Attachment Systems in Mandibular Single Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Sedky Abd El-lateef, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: single implant overdenture
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Patient Satisfaction; Edentulous Mandible
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessor of 1ry outcome, statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ball and socket attachment (Active Comparator): mandibular single implant overdenture retained by ball and socket attachment
  Interventions: Other: ball and socket attachment
- locator attachment (Experimental): mandibular single implant overdenture retained by locator attachment
  Interventions: Other: locator attachment

INTERVENTIONS:
Other: locator attachment — mandibular single implant overdenture retained by locator attachment
  Arms: locator attachment
Other: ball and socket attachment — mandibular single implant overdenture retained by ball and socket attachment
  Arms: ball and socket attachment

SUMMARY:
to compare locator attachment to ball attachment in retaining mandibular single implant overdenture in terms of patient satisfaction and retention

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous patient
2. Patients having enough bone for an implant length of at least 10 mm
3. Sufficient inter-arch space to accommodate the denture & the attachment
4. No apparent Skeletal mal-relation
5. No intraoral soft and hard tissue pathology
6. No systemic condition that contraindicate implant placement

Exclusion Criteria:

1. Drug or alcohol abuse
2. Smokers
3. A health condition precluding surgery,
4. Logistic or physical reasons that could affect follow-up,
5. Psychiatric problems
6. Medically compromised patients & those with neuromascular disorders
7. Disorders to the implant area related to a history of radiation therapy to the head and neck, neoplasia, or bone augmentation to the implant site.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | baseline, 1month, 6 months, 1 and 3 years
  Patient satisfaction will be measured using a valid and reliable questionnaire which is Patient satisfaction with lower removable denture questionnaire SLRD-Q. likert scale ranges from very good (1) to good (2), neither good nor bad (3), bad (4), and extremely bad (5)

SECONDARY OUTCOMES:
Retention | baseline, 1 month, 3 and 6 months
  Measuring device: Force meter Measuring unit: Newton/cm2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt